CLINICAL TRIAL: NCT06974396
Title: Comparative Evaluation of the Performance of Different Thromboplastin Reagents on Prothrombin Time and Factorial Assays in Situations of Isolated Extrinsic Pathway Factor Deficiency or Liver Damage
Brief Title: Comparative Evaluation of the Performance of Different Thromboplastin Reagents on Prothrombin Time in Situations of Isolated Extrinsic Pathway Factor Deficiency or Liver Damage
Acronym: RHEOMICS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9696
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Hemorrhagic Disorders
MeSH Terms: conditions — Hemorrhagic Disorders | interventions — Prothrombin Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolated extrinsic pathway factor deficiency (Other): Patients with an isolated extrinsic pathway factor deficiency (acquired or congenital) : II or V or VII or X
  Interventions: Biological: Prothrombin time
- Hepatocellular insufficiency with coagulopathy (Other): Patients with an hepatocellular insufficiency generally associated with coagulopathy (with an intensity proportional to the degree of hepatic impairment).
  Interventions: Biological: Prothrombin time

INTERVENTIONS:
Biological: Prothrombin time — Comparison of prothrombin time results obtained with the different thromboplastins reagent for subgroup (extrinsic pathway factor and for those with hepatocellular insufficiency) by a regression line and a Bland-Altman representation.
  Comparison of extrinsic pathway factor assays obtained with the different thromboplastins reagent for each subgroup by a regression line and a Bland-Altman representation.
  Evaluation and determination of the sensitivity of the prothrombin time according to the activity rate obtained for each factor (for each reagent).

SUMMARY:
Primary purpose :

Compare the sensitivity of several thromboplastin reagents of various origins to prothrombin time and factor II, V, VII and X assays in two different populations of patients :

* Patients with an isolated extrinsic pathway deficiency (acquired or congenital) of factor II or V or VII or X.
* Patients with an hepatocellular insufficiency generally associated with coagulopathy (with an intensity proportional to the degree of hepatic impairment).

Results of this work should improve knowledge of sensitivity of the screening test represented by the prothrombin time, depending on the origin of thromboplastin reagent used, in relation with coagulopathies mentioned above, as well as the performance of factors II, V, VII, X assays. This work would help to choice of the most suitable reagent for the needs of each hemostasis laboratory/center.

ELIGIBILITY:
Inclusion Criteria:

* Plasma samples from patients addressed to the laboratory of the Strasbourg University Hospital (Strasbourg France) collected and anonymized after completion of the routine testing.
* Patient with an isolated or combined extrinsic pathway factor deficiency (factor II, V, VII, X).

Exclusion Criteria:

* Patient treated with an oral anticoagulant treatment.
* Patient treated with a parenteral anticoagulant treatment (apart from therapeutic dosages of unfractionated heparin and low molecular weight heparin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the sensitivity of several thromboplastin reagents of different origins (animal, human synthetic recombinant and human placental extraction) on prothrombin time and factor II, V, VII and X assays. | Plasma samples were frozen at -80°C within 3 hours of collection and were serially analyzed few weeks later by thawing at 37°C within 2 hours after thawing.

IPD SHARING:
Plan to Share IPD: No